CLINICAL TRIAL: NCT04837820
Title: Effect and Mechanism of Acupuncture for Cancer-related Cognitive Difficulties (ENHANCE)
Brief Title: The Effect of Acupuncture on Cancer-Related Cognitive Difficulties
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20-124
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer
Keywords: Acupuncture; Cancer-Related Cognitive Difficulties; 20-124
MeSH Terms: conditions — Breast Neoplasms | interventions — Acupuncture Therapy; Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: 3-arm, parallel, randomized controlled trial comparing acupuncture vs. sham acupuncture vs. wait-list control.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acupuncture (Experimental): The intervention will consist of 10 acupuncture sessions over 10 weeks using the standardized, semi-fixed protocol.
  Interventions: Procedure: Acupuncture; Other: Questionnaires
- Sham Acupuncture (SA) (Placebo Comparator): The intervention will consist of 10 acupuncture sessions over 10 weeks using the standardized, semi-fixed protocol.
  Interventions: Procedure: Sham Acupuncture; Other: Questionnaires
- Wait-List Control (Experimental): During the 26-week waiting period, the CRC will contact patients in the WLC group at the same frequency as the acupuncture groups with respect to data collection. Patients in the WLC group will continue to receive their standard medical care as prescribed by their oncologists/primary care physicians. WLC patients will be compensated with real acupuncture treatments after Week 26 (end of study).
  Interventions: Other: Wait-List Control (WLC); Other: Questionnaires

INTERVENTIONS:
Procedure: Acupuncture — Each participant will receive 10 treatments of acupuncture (real or sham) over the course of 10 weeks (i.e. one treatment a week) with a +/- 14-day window.
  Arms: Acupuncture
Procedure: Sham Acupuncture — Each participant will receive 10 treatments of acupuncture (real or sham) over the course of 10 weeks (i.e. one treatment a week) with a +/- 14-day window.
  Arms: Sham Acupuncture (SA)
Other: Wait-List Control (WLC) — Patients in the WLC group will continue to receive their standard medical care as prescribed by their oncologists/primary care physicians.
  Arms: Wait-List Control
Other: Questionnaires — Will follow patients for 26 weeks from baseline and collect assessments at baseline and Weeks 0, 10, and 26. Average time to complete the surveys is 30 minutes, which has been judged to be acceptable with minimal missing data; 20 minutes of these 30 minutes will be completed during the neurocognitive battery. Patients will complete PROs online using Research Electronic Data Capture (REDCap) or over the phone with the CRC. Biospecimens will be collected in person at assessment visits. The neurocognitive battery will be administered remotely.

SUMMARY:
The purpose of this study is to test whether acupuncture can improve cognitive difficulties and insomnia in survivors of breast cancer. Researchers will compare the effects of real acupuncture with those of placebo acupuncture and wait-list acupuncture. This study will also look at insomnia's link to cognitive difficulties.

All study participants (receiving real acupuncture, placebo acupuncture, or wait-list acupuncture) will complete study questionnaires and/or have cognitive testing at Weeks 0, 4, 10, 14 and 26. After the Week 26 visit, your participation in this study will end. If you are assigned to receive placebo acupuncture or wait-list acupuncture, you will have the option of receiving up to 10 real acupuncture treatments within the six months after the study finishes.

ELIGIBILITY:
Inclusion Criteria:

* English-proficient adult women with a history of stage 0, I, II, or III breast cancer
* Free of oncologic disease by clinical examination or history
* Moderate or greater CRCD as indicated by a score of "quite a bit" or "very much" on at least one of the two items that specifically assess concentration and memory on the EORTC QLQ-C30 (version 3.0)
* Report that cognitive functions worsened since cancer diagnosis by replying "Yes" to all 3 questions

  * Do you think or feel that your memory or mental ability has gotten worse since your cancer diagnosis?
  * Do you think your mind isn't as sharp now as it was before your cancer diagnosis?
  * Do you feel like these problems have made it harder to function on your job or take care of things around the home?
* Presence of insomnia symptoms as indicated by a score ≥8 on the ISI134
* Willing to adhere to all study-related procedures, including randomization to one of the 3 possible choices: acupuncture, sham acupuncture, or wait-list control

Exclusion Criteria:

* Metastatic breast cancer (stage IV)
* Less than 1 month since completion of surgery, chemotherapy or radiation therapy
* Greater than 10 years since most recent breast cancer diagnosis
* Use of acupuncture for sleep or cognitive symptom management within the past 3 months
* Diagnosis of Alzheimer's disease, vascular dementia, Parkinson disease, or other organic brain disorder
* Score of >10 indicative of overt dementia on the Blessed Orientation-Memory-Concentration (BOMC)135
* Primary psychiatric disorder not in remission
* As per medical record or self-report, history of stroke or head injury requiring visit to the emergency room or hospitalization, with confirmed structural lesion on neuroimaging, persistent cognitive difficulties impacting work or daily life, or required cognitive rehabilitation.
* Pre-existing, uncorrectable visual or auditory impairment that would preclude ability to complete the assessments
* Initiation or change in hormonal or targeted therapy within the past 4 weeks
* Plans to initiate or change hormonal or targeted therapy in the coming 8 weeks
* Altered dose of somnogenic medication (e.g. hypnotics, sedatives, antidepressants) in past 8 weeks
* Enrolled or plans to enroll on another MSK neurocognitive study
* Unable to provide informed consent for himself/herself

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast Cancer
Enrollment: 270 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
cognitive difficulties | 26 weeks
  measured by the Functional Assessment of Cancer Therapy - Cognitive Function (FACT-Cog) instrument. FACT-Cog is a 37-item questionnaire with 4 subscales: perceived cognitive difficulties, impact on quality of life, comments from others, and perceived cognitive abilities. The FACT-Cog perceived cognitive impairment subscale (Cronbach's α 0.94) will be the primary outcome for the study. A subscale score is calculated by summing the 18 items of the subscale. The subscale score ranges from 0 to 72.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Mao, MD, MSCE, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk- Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

DOCUMENTS (1):
  • Informed Consent Form (2024-02-20): https://cdn.clinicaltrials.gov/large-docs/20/NCT04837820/ICF_000.pdf